CLINICAL TRIAL: NCT01775813
Title: Combined Influence of Puberty and Obesity on Insulin Resistance in Adolescents
Brief Title: The Health Influences of Puberty (HIP) Study
Acronym: HIP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Diabetes Association (Other); National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 07-0988; Protocol 914 (Other: Children's Hospital Colorado); 1-11-JF-23 (Other Grant/Funding Number: American Diabetes Association); 5K12HD057022 (NIH)
Record Dates: First submitted 2012-10-05; First posted 2013-01-25 (Estimated); Results first posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Obesity; Insulin Resistance; Gonadal Dysfunction; Type 2 Diabetes
Keywords: Insulin resistance; Puberty; Obesity; Hypogonadism; Gonadal dysfunction; Metformin
MeSH Terms: conditions — Obesity; Insulin Resistance; Gonadal Disorders; Diabetes Mellitus, Type 2; Hypogonadism | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Obese metformin arm (Experimental): Double-blinded placebo-controlled trial of metformin during puberty, treatment arm Dosage form: Metformin 1000 mg tablets Dosage: 1000 mg by mouth twice daily Duration: From early puberty (Tanner 2-3) until puberty completion (Tanner 5), approximately 3 years
  Interventions: Drug: Metformin
- Obese placebo arm (Placebo Comparator): Double-blinded placebo-controlled trial of metformin during puberty, placebo arm Dosage form: Placebo stamped to match 1000 mg metformin tablets Placebo comparator: Stamped placebo pill matching metformin dose Dosage: 1000 mg by mouth twice daily Duration: From early puberty (Tanner 2-3) until puberty completion (Tanner 5), approximately 3 years
  Interventions: Drug: Placebo
- Obese - NT (No Intervention): Comparator group for the observational comparison of metabolic changes in youth with normal weight and obesity as they progress through puberty.
  Duration: From early puberty (Tanner 2-3) until puberty completion (Tanner 5), approximately 3 years
- Normal weight (No Intervention): Comparator group for the observational comparison of metabolic changes in youth with normal weight and obesity as they progress through puberty.
  Duration: From early puberty (Tanner 2-3) until puberty completion (Tanner 5), approximately 3 years

INTERVENTIONS:
Drug: Metformin — After randomization, the study drug (metformin or placebo) is gradually titrated to full dose of 1000 mg BID (or to maximum tolerated, at least 500 mg BID) over a period of 4 weeks to minimize adverse gastrointestinal effects. Participants are seen every three months to measure compliance and dispense new study drug. Every 6 months, they also have a physical examination in order to determine puberty staging. Study measurements (IVGTT, bloodwork, DXA) are performed at Tanner 4 puberty and Tanner 5 (puberty completion), at which time the study drug is stopped. Study measurements will be performed again 6 months after study drug is completed to assess if effects are persistent after study drug is stopped. During the treatment period, all participants receive standard lifestyle counseling.
  Other Names: Glucophage; Glumetza; Fortamet; Riomet
  Arms: Obese metformin arm
Drug: Placebo — Stamped placebo pill to look like the 1000 mg metformin pill Dosage: 1 pill taken orally twice daily Duration: From early puberty (Tanner 3-4) until puberty completion (Tanner 5), approximately 3 years
  Arms: Obese placebo arm

SUMMARY:
The Health Influences of Puberty (HIP) Study is designed to explore the relationships between puberty and the onset of type 2 diabetes in adolescents. The results of this study will help us better understand how to prevent type 2 diabetes in these youth. Children go through many changes during puberty, including important hormonal and behavioral alterations. Among these changes, it has long been known that, during puberty, insulin does not work as well as it does before and after puberty. This is called physiologic insulin resistance. In healthy children, this does not cause diabetes or affect blood sugar in any way because the body is able to compensate by making more insulin. Indeed, this is thought to be an important part of the adolescent growth spurt. However, in some children with increased risk for developing type 2 diabetes due to obesity and genetics, the worsening insulin resistance of puberty cannot be compensated for and these youth get diabetes early. The investigators believe this is because type 2 diabetes is rarely, if ever, seen before puberty begins, and the peak of diabetes onset in adolescents occurs at the time of the worst insulin resistance. This specific research project has two goals: 1. To examine effects of obesity on how well the body's insulin works during puberty, and 2. To see if treatment of obese children during this critical period of puberty with a medication that improves insulin resistance (metformin) will help prevent early onset type 2 diabetes.

DETAILED DESCRIPTION:
Specific Aims:

Pediatric insulin resistance and related disorders, such as type 2 diabetes mellitus (T2DM), are increasing in prevalence, and portend significant end-organ and cardiovascular morbidity and mortality. Thus, measures aimed at understanding its causes and preventing its onset are critical. The physiologic decrease in insulin sensitivity in all adolescents during puberty is well-established. It is also known that obese adolescents start out less insulin sensitive at the onset of puberty than lean adolescents, and that their insulin sensitivity worsens as puberty progresses. While there are both longitudinal and cross-sectional data confirming the natural recovery of pre-pubertal insulin sensitivity in normal weight adolescents after puberty is completed, it is unknown whether obese adolescents recover their pre-pubertal insulin sensitivity. Failure to regain pre-pubertal insulin sensitivity at the end of puberty, and failure of compensatory insulin secretion, may accelerate progression from obesity to insulin resistance to T2DM in at-risk youth and contribute to long-term cardiovascular risk.

In addition, obesity and insulin resistance are associated with earlier onset of puberty and premature adrenarche in females. Insulin resistance also contributes to the gonadal dysfunction of polycystic ovarian disease in fully pubertal females and is associated with hypogonadism in older adult males. Little is known about effects of obesity and insulin resistance on gonadal function in young males. However, persistent metabolic changes at the end of puberty may contribute to gonadal dysfunction in obese youth. Currently, there are few longitudinal studies in either sex that evaluate the interactions among obesity, insulin resistance and gonadal function during puberty.

The investigators' long-term goal is to better understand the metabolic changes that occur during puberty, their underlying mechanisms, and their potential contribution to adult disease. The overall aim is to evaluate the effects of obesity on the evolution of insulin sensitivity and gonadal function during puberty. In addition, because improvement in insulin action during puberty may slow β-cell deterioration, the investigators will evaluate whether compensatory insulin secretion is also affected in obese adolescents and whether treatment with metformin improves β-cell response.

HYPOTHESES:

1. Obese adolescents will show decreased improvement in insulin sensitivity from Tanner stage 2/3 to Tanner 5 when compared with lean counterparts.
2. Obese adolescents treated with metformin will have greater improvement in insulin sensitivity from Tanner stage 2/3 to Tanner 5 vs. those treated with placebo. (See hypothesis schematics below)

To test these hypotheses, we propose to address the following Specific Aims:

SPECIFIC AIM 1 (Observational Arm):

1. To compare longitudinal changes in insulin sensitivity and secretion and their correlates in obese and normal weight adolescents during puberty.

   1. Primary outcome: Change in insulin sensitivity (Si), as measured by frequently sampled intravenous glucose tolerance test (IVGTT), from early puberty to puberty completion in obese and normal weight adolescents.
   2. Secondary outcomes: Change in insulin secretion (AIR) and disposition index (DI) as measured by IVGTT, body composition, fat distribution, markers of gonadal function, and inflammatory markers over time in these groups.

   SPECIFIC AIM 2 (Treatment Arm):
2. To compare longitudinal changes in insulin sensitivity and secretion and their correlates in obese adolescents treated with metformin or placebo during puberty.

   1. Primary outcome: Change in Si from early puberty to puberty completion in obese controls and obese adolescents treated with metformin.
   2. Secondary outcome: Change in AIR and DI, body composition, fat distribution, markers of gonadal function, and inflammatory markers over time in these groups.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 95th percentile
* At least Tanner 2, but no more than Tanner 3
* Age ≥ 9 years
* Absence of impaired glucose tolerance (IGT), impaired fasting glucose (IFG) or Type 2 diabetes mellitus (T2DM)

Exclusion Criteria:

* Presence of T2DM, IGT or IFG
* Any disorder or medication known to effect glucose tolerance;
* Hypertension or hyperlipidemia requiring pharmacological intervention;
* Weight >300lbs. due to limits of imaging tables.
* Chronic illness

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Kelsey, MD, MS, Principal Investigator — University of Colorado Denver/Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

REFERENCES:
- [Derived] Kelsey MM, Hilkin A, Pyle L, Severn C, Utzschneider K, Van Pelt RE, Zeitler PS, Nadeau KJ. Two-Year Treatment With Metformin During Puberty Does Not Preserve beta-Cell Function in Youth With Obesity. J Clin Endocrinol Metab. 2021 Jun 16;106(7):e2622-e2632. doi: 10.1210/clinem/dgab170. PMID 33728428
- [Derived] Kelsey MM, Pyle L, Hilkin A, Severn CD, Utzschneider K, Van Pelt RE, Nadeau KJ, Zeitler PS. The Impact of Obesity On Insulin Sensitivity and Secretion During Pubertal Progression: A Longitudinal Study. J Clin Endocrinol Metab. 2020 May 1;105(5):e2061-8. doi: 10.1210/clinem/dgaa043. PMID 31996919

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Weight: Normal Weight by BMI. No treatment.
- Obese - NT: Obese by BMI. These participants were not prescribed any intervention (Non-treated).
- Obese - Placebo: Dosage form: Stamped placebo pill to look like the 1000 mg metformin pill Dosage: 1 pill taken orally twice daily Duration: From early puberty (Tanner 3-4) until puberty completion (Tanner 5), approximately 3 years
- Obese - Metformin: Dosage form: Metformin 1000 mg tablets Dosage: 1000 mg by mouth twice daily Duration: From early puberty (Tanner 3-4) until puberty completion (Tanner 5), approximately 3 years
Period: Overall Study
Arm/Group | Normal Weight | Obese - NT | Obese - Placebo | Obese - Metformin
Started (Patients that had data collected at Study Visit 1 (1st IVGTT)) | 47 | 13 | 24 | 20
Study Visit 2 (Tanner 4) | 36 | 4 | 11 | 11
Study Visit 3 (Tanner 5) | 34 | 8 | 12 | 11
Study Visit 4 (Post-Puberty) | 10 | 0 | 13 | 11
Completed (Patients that completed Study Visit 3 (Primary Outcome)) | 34 | 8 | 12 | 11
Not Completed | 13 | 5 | 12 | 9

BASELINE CHARACTERISTICS:
Population: Both the Obese - NT participants and Obese - Placebo participants were included in the "observational arm" of the study. Thus, this arm was a comparison between youth with normal weight and untreated and youth with obesity who were either a) untreated or b) treated with placebo
Groups:
- Obese - NT: Obese by BMI. Participants were not taking metformin or placebo
- Total: Total of all reporting groups
Arm/Group | Normal Weight | Obese - NT | Obese - Placebo | Obese - Metformin | Total
Number analyzed (Participants) | 47 | 13 | 24 | 20 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.070 (1.513) | 11.274 (1.138) | 11.146 (1.088) | 11.863 (1.562) | 11.754 (1.437)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 6 | 17 | 9 | 54
  Male | 25 | 7 | 7 | 11 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 12 | 7 | 19 | 16 | 54
  Non-Hispanic White | 23 | 4 | 2 | 1 | 30
  Black | 8 | 1 | 2 | 2 | 13
  Asian | 3 | 0 | 0 | 0 | 3
  Other | 1 | 1 | 1 | 0 | 3
  Native American | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 47 | 13 | 24 | 20 | 104

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: As measured by in intravenous glucose tolerance test (IVGTT) as calculated by Bergman's minimal model. Higher numbers indicate a better outcome. Patients are randomized to receive metformin or placebo at Tanner stage 2-3 of puberty. They are reassessed at Tanner 4 and again at Tanner 5. At that point, the treatment is stopped and they are reassessed 6 months after stopping treatment to see if effects of treatment persist.
Time Frame: Baseline, Tanner (puberty) stage 4-average 1.5 years from baseline, Tanner (puberty) stage 5-average 2.5 yrs from baseline, 6 mos post-treatment-average 3 yrs from baseline
Population: 24 participants analyzed in the Obese NT Placebo group are also analyzed in the Obese Placebo group.
Measure: Mean (Standard Deviation); unit: x10-4/min-1/mIU/mL
Groups:
- Obese - NT: Obese by BMI. These participants were not assigned an intervention (non-treated).
Arm/Group | Normal Weight | Obese - NT | Obese - Placebo | Obese - Metformin
Number analyzed (Participants) | 47 | 37 | 24 | 20
x10-4/min-1/mIU/mL
  Baseline | 8.559 (5.755) | 3.425 (4.197) | 3.756 (4.970) | 2.985 (2.656)
  Tanner 4 | 6.661 (4.418) | 1.995 (0.959) | 1.868 (1.102) | 2.873 (2.155)
  Tanner 5 | 6.438 (3.835) | 2.082 (1.764) | 2.383 (2.056) | 2.990 (3.038)
  Post-Puberty | NA (NA) — Not Measured | NA (NA) — Not Measured | 3.017 (3.449) | 2.182 (2.353)

2. Secondary Outcome: Insulin Secretion (Acute Insulin Response to Glucose, AIRg)
Description: As measured by IVGTT as calculated by Bergman's minimal model. Higher numbers indicate a better outcome. Please see primary outcome for more detail about timing of measurement.
Time Frame: as for outcome 1
Population: 24 participants analyzed in the Obese NT Placebo group are also analyzed in the Obese Placebo group.
Measure: Mean (Standard Deviation); unit: µIU/mL
Groups:
- Obese - NT/Placebo: Obese by BMI. Mixture of non treated and placebo treated patients.
Arm/Group | Normal Weight | Obese - NT/Placebo | Obese - Placebo | Obese - Metformin
Number analyzed (Participants) | 47 | 37 | 24 | 20
µIU/mL
  Baseline | 583.535 (432.753) | 1877.895 (1052.328) | 1858.16 (1079.128) | 2368.931 (1616.348)
  Tanner 4 | 783.191 (623.946) | 1951.323 (1035.697) | 1996.867 (1215.017) | 2157.349 (1099.876)
  Tanner 5 | 680.858 (572.884) | 2103.309 (1505.040) | 2013.628 (1417.407) | 1804.026 (761.849)
  Post-Puberty | NA (NA) — Not Measured | NA (NA) — Not Measured | 1943.542 (1353.036) | 1667.713 (917.270)

3. Secondary Outcome: Disposition Index
Description: Please see primary outcome for more detail about timing of measurement. Disposition index is measured via (IVGTT) as calculated by Bergman's minimal model. Higher numbers indicate a better outcome. It reflects the product of outcome measures 1 and 2 (Si x AIRg).
Time Frame: as for outcome 1
Population: 24 participants analyzed in the Obese NT Placebo group are also analyzed in the Obese Placebo group.
Measure: Mean (Standard Deviation); unit: x10-4/min-1
Arm/Group | Normal Weight | Obese - NT/Placebo | Obese - Placebo | Obese - Metformin
Number analyzed (Participants) | 47 | 37 | 24 | 20
x10-4/min-1
  Baseline | 3750.463 (1625.015) | 4195.921 (1743.345) | 4286.209 (1966.920) | 4438.821 (2420.123)
  Tanner 4 | 3706.940 (1972.563) | 3269.039 (1500.261) | 2897.689 (1553.948) | 5046.218 (2858.784)
  Tanner 5 | 3234.061 (2474.754) | 2897.244 (1547.515) | 3194.773 (1918.812) | 3537.273 (768.858)
  Post-Puberty | NA (NA) — Not Measured | NA (NA) — Not Measured | 3627.762 (2375.166) | 2539.933 (1393.267)

4. Secondary Outcome: Low Density Lipoprotein
Description: Please see primary outcome for more detail about timing of measurement.
Time Frame: as for outcome 1
Population: 24 participants analyzed in the Obese NT Placebo group are also analyzed in the Obese Placebo group.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Normal Weight | Obese - NT/Placebo | Obese - Placebo | Obese - Metformin
Number analyzed (Participants) | 47 | 37 | 24 | 20
mg/dl
  Baseline | 79.488 (22.691) | 86.533 (22.543) | 88.583 (23.824) | 83.779 (25.029)
  Tanner 4 | 75.367 (15.852) | 96.636 (19.464) | 96.636 (19.464) | 81.818 (24.677)
  Tanner 5 | 78.485 (20.520) | 96.222 (24.422) | 97.667 (27.655) | 75.000 (27.799)
  Post-Puberty | NA (NA) — Not Measured | NA (NA) — Not Measured | 103.154 (26.620) | 86.545 (28.507)

5. Secondary Outcome: Insulin-like Growth Factor 1
Description: IGF-1 measured in serum at each time point
Time Frame: Baseline, Tanner (puberty) stage 4-average 1.5 years from baseline, Tanner (puberty) stage 5-average 2.5 yrs from baseline
Population: 24 participants analyzed in the Obese NT Placebo group are also analyzed in the Obese Placebo group.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Normal Weight | Obese - NT/Placebo | Obese - Placebo | Obese - Metformin
Number analyzed (Participants) | 47 | 37 | 24 | 20
ng/ml
  Baseline | 313.500 (103.339) | 262.278 (91.924) | 243.042 (85.040) | 281.700 (86.014)
  Tanner 4 | 405.389 (116.845) | 370.800 (89.816) | 380.273 (77.040) | 410.300 (116.467)
  Tanner 5 | 398.000 (97.117) | 389.800 (116.087) | 351.833 (74.909) | 404.800 (88.745)
  Post-Puberty | NA (NA) — Not Measured | NA (NA) — Not Measured | 319.692 (93.694) | 395.818 (114.417)

6. Secondary Outcome: Total Testosterone
Description: Testosterone measured in serum at each time point
Time Frame: as for outcome 5
Population: 24 participants analyzed in the Obese NT Placebo group are also analyzed in the Obese Placebo group.
Measure: Mean (Standard Deviation); unit: ng/dl
Arm/Group | Normal Weight | Obese - NT/Placebo | Obese - Placebo | Obese - Metformin
Number analyzed (Participants) | 47 | 37 | 24 | 20
ng/dl
  Baseline | 108.625 (135.377) | 35.278 (28.375) | 30.125 (20.422) | 41.050 (32.705)
  Tanner 4 | 145.972 (159.866) | 87.933 (103.902) | 89.364 (105.331) | 121.727 (113.418)
  Tanner 5 | 235.559 (235.224) | 158.300 (234.056) | 165.750 (282.171) | 117.909 (132.301)
  Post-Puberty | NA (NA) — Not Measured | NA (NA) — Not Measured | 152.692 (168.109) | 150.727 (161.357)

7. Secondary Outcome: Estradiol
Description: Estradiol measured in serum at each time point
Time Frame: as for outcome 5
Population: 24 participants analyzed in the Obese NT Placebo group are also analyzed in the Obese Placebo group.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Normal Weight | Obese - NT/Placebo | Obese - Placebo | Obese - Metformin
Number analyzed (Participants) | 47 | 37 | 24 | 20
pg/mL
  Baseline | 22.375 (34.068) | 15.722 (7.756) | 15.833 (7.738) | 14.750 (6.695)
  Tanner 4 | 50.583 (70.888) | 35.867 (49.693) | 44.545 (56.077) | 23.364 (14.123)
  Tanner 5 | 57.382 (79.251) | 42.800 (38.324) | 48.833 (47.610) | 48.000 (29.192)
  Post-Puberty | NA (NA) — Not Measured | NA (NA) — Not Measured | 70.923 (91.316) | 69.636 (85.940)

8. Secondary Outcome: Sex Hormone Binding Globulin
Description: SHBG measured in serum at each time point
Time Frame: as for outcome 5
Population: 24 participants analyzed in the Obese NT Placebo group are also analyzed in the Obese Placebo group.
Measure: Mean (Standard Deviation); unit: nmol/l
Arm/Group | Normal Weight | Obese - NT/Placebo | Obese - Placebo | Obese - Metformin
Number analyzed (Participants) | 47 | 37 | 24 | 20
nmol/l
  Baseline | 61.958 (21.680) | 20.417 (8.310) | 18.958 (6.805) | 17.550 (8.451)
  Tanner 4 | 50.417 (24.098) | 17.200 (7.580) | 16.364 (6.742) | 19.545 (14.348)
  Tanner 5 | 43.500 (15.498) | 16.250 (5.581) | 15.750 (6.468) | 16.455 (8.825)
  Post-Puberty | NA (NA) — Not Measured | NA (NA) — Not Measured | 15.538 (4.409) | 17.273 (10.640)

9. Secondary Outcome: Dehydroepiandrosterone Sulfate
Description: DHEA-S measured in serum at each time point
Time Frame: as for outcome 5
Measure: Mean (Standard Deviation); unit: mcg/dl
Arm/Group | Normal Weight | Obese - NT/Placebo | Obese - Placebo | Obese - Metformin
Number analyzed (Participants) | 47 | 37 | 24 | 20
mcg/dl
  Baseline | 90.146 (60.522) | 96.750 (63.592) | 91.167 (60.501) | 107.600 (64.722)
  Tanner 4 | 101.889 (62.016) | 101.533 (67.038) | 116.182 (71.822) | 129.545 (69.398)
  Tanner 5 | 130.206 (69.229) | 137.250 (74.248) | 137.083 (86.885) | 145.818 (66.535)
  Post-Puberty | NA (NA) — Not Measured | NA (NA) — Not Measured | 132.154 (68.295) | 176.818 (110.840)

10. Secondary Outcome: High Sensitivity C-reactive Protein
Description: hsCRP measured in serum at each time point
Time Frame: as for outcome 5
Population: 24 participants analyzed in the Obese NT Placebo group are also analyzed in the Obese Placebo group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Normal Weight | Obese - NT/Placebo | Obese - Placebo | Obese - Metformin
Number analyzed (Participants) | 47 | 37 | 24 | 20
units on a scale
  Baseline | 1.001 (2.604) | 2.523 (2.644) | 3.117 (3.060) | 3.962 (3.608)
  Tanner 4 | 0.305 (0.631) | 4.530 (5.034) | 4.357 (5.661) | 1.841 (1.494)
  Tanner 5 | 1.015 (3.265) | 3.331 (3.814) | 3.985 (4.681) | 0.961 (0.915)
  Post-Puberty | NA (NA) — Not Measured | NA (NA) — Not Measured | 3.958 (3.510) | 2.667 (4.647)

11. Secondary Outcome: Aspartate Aminotransferase (AST)
Description: AST measured in serum at each time point
Time Frame: as for outcome 5
Population: 24 participants analyzed in the Obese NT Placebo group are also analyzed in the Obese Placebo group.
Measure: Mean (Standard Deviation); unit: international units per liter
Arm/Group | Normal Weight | Obese - NT/Placebo | Obese - Placebo | Obese - Metformin
Number analyzed (Participants) | 47 | 37 | 24 | 20
international units per liter
  Baseline | 42.174 (14.685) | 41.250 (18.130) | 43.542 (20.156) | 54.150 (28.117)
  Tanner 4 | 35.706 (11.202) | 44.429 (25.621) | 43.636 (26.070) | 40.273 (14.065)
  Tanner 5 | 33.364 (11.811) | 36.650 (17.458) | 42.333 (20.331) | 34.091 (11.122)
  Post-Puberty | NA (NA) — Not Measured | NA (NA) — Not Measured | 39.077 (21.278) | 36.273 (17.396)

12. Secondary Outcome: Alanine Transaminase (ALT)
Description: ALT measured in serum at each time point
Time Frame: Baseline (Tanner 2-3), Tanner 4, Tanner 5
Population: 24 participants analyzed in the Obese NT Placebo group are also analyzed in the Obese Placebo group.
Measure: Mean (Standard Deviation); unit: international units per liter
Arm/Group | Normal Weight | Obese - NT/Placebo | Obese - Placebo | Obese - Metformin
Number analyzed (Participants) | 47 | 37 | 24 | 20
international units per liter
  Baseline | 25.022 (9.556) | 35.194 (22.132) | 41.125 (24.552) | 52.400 (50.296)
  Tanner 4 | 27.059 (7.671) | 44.571 (40.839) | 51.182 (43.829) | 42.545 (18.753)
  Tanner 5 | 26.121 (6.859) | 38.650 (23.089) | 47.500 (25.995) | 39.636 (17.328)
  Post-Puberty | NA (NA) — Not Measured | NA (NA) — Not Measured | 50.231 (36.967) | 45.000 (30.864)

13. Secondary Outcome: Change in Urinary Luteinizing Hormone
Description: LH measured in an overnight urine sample at time points below
Time Frame: Baseline, every 6 months during the trial, Final visit (average 3 yrs after baseline)
Population: 24 participants analyzed in the Obese NT Placebo group are also analyzed in the Obese Placebo group.
Measure: Mean (Standard Deviation); unit: international units per liter
Arm/Group | Normal Weight | Obese - NT/Placebo | Obese - Placebo | Obese - Metformin
Number analyzed (Participants) | 47 | 37 | 24 | 20
international units per liter
  Tanner 2/3 | 3.849 (4.530) | 2.257 (2.186) | 2.257 (2.186) | 3.809 (3.667)
  Tanner 4 | 4.518 (8.496) | 3.310 (3.793) | 3.310 (3.793) | 3.729 (4.036)
  Tanner 5 | 4.494 (7.616) | 2.014 (1.442) | 2.014 (1.442) | 8.993 (14.725)
  Post-Puberty | NA (NA) — Not Measured | 5.373 (11.363) | 5.373 (11.363) | 30.861 (62.387)

14. Secondary Outcome: Change in Urinary Follicle-stimulating Hormone
Description: FSH measured in overnight urine sample at time points below
Time Frame: Baseline, every 6 months during the trial, Final visit-average 3 yrs after baseline
Population: 24 participants analyzed in the Obese NT Placebo group are also analyzed in the Obese Placebo group.
Measure: Mean (Standard Deviation); unit: international units per milliliter (IU/m
Arm/Group | Normal Weight | Obese - NT/Placebo | Obese - Placebo | Obese - Metformin
Number analyzed (Participants) | 47 | 37 | 24 | 20
international units per milliliter (IU/m
  Tanner 2/3 | 3.911 (5.590) | 3.837 (4.264) | 3.837 (4.264) | 3.615 (4.356)
  Tanner 4 | 2.555 (2.541) | 4.874 (3.586) | 4.874 (3.586) | 3.162 (2.686)
  Tanner 5 | 6.540 (9.360) | 4.093 (3.962) | 4.093 (3.962) | 3.213 (3.323)
  Post-Puberty | NA (NA) — Not Measured | 5.993 (6.429) | 5.993 (6.429) | 3.911 (2.689)

15. Secondary Outcome: Change in Urinary Estradiol Metabolites
Description: estradiol metabolite (E1c) measured in an overnight urine sample at each time point
Time Frame: Baseline, every 6 months during the trial, Final visit-average 3 yrs after baseline
Population: 24 participants analyzed in the Obese NT Placebo group are also analyzed in the Obese Placebo group.
Measure: Mean (Standard Deviation); unit: ng/mgCr
Arm/Group | Normal Weight | Obese - NT/Placebo | Obese - Placebo | Obese - Metformin
Number analyzed (Participants) | 47 | 37 | 24 | 20
ng/mgCr
  Tanner 2/3 | 7.711 (22.531) | 17.353 (17.214) | 17.353 (17.214) | 28.451 (26.082)
  Tanner 4 | 22.919 (37.835) | 8.584 (9.932) | 8.584 (9.932) | 37.722 (34.648)
  Tanner 5 | 41.036 (78.160) | 7.825 (2.586) | 7.825 (2.586) | 71.546 (77.343)
  Post-Puberty | NA (NA) — Not Measured | 26.402 (38.299) | 26.402 (38.299) | 30.883 (33.674)

16. Secondary Outcome: Hemoglobin A1c
Description: HbA1c measured by HPLC at time points below
Time Frame: as for outcome 5
Population: 24 participants analyzed in the Obese NT Placebo group are also analyzed in the Obese Placebo group.
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Normal Weight | Obese - NT/Placebo | Obese - Placebo | Obese - Metformin
Number analyzed (Participants) | 47 | 37 | 24 | 20
mmol/mol
  Baseline | 5.139 (0.250) | 5.336 (0.488) | 5.336 (0.488) | 5.400 (0.286)
  Tanner 4 | 5.200 (0.260) | 5.627 (0.531) | 5.627 (0.531) | 5.570 (0.250)
  Tanner 5 | 5.233 (0.293) | 5.476 (0.360) | 5.500 (0.398) | 5.473 (0.552)
  Post-Puberty | NA (NA) — Not Measured | NA (NA) — Not Measured | 5.515 (0.519) | 5.691 (0.929)

17. Secondary Outcome: Leptin
Description: Leptin measured in serum at time points below
Time Frame: as for outcome 5
Population: 24 participants analyzed in the Obese NT Placebo group are also analyzed in the Obese Placebo group.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Normal Weight | Obese - NT/Placebo | Obese - Placebo | Obese - Metformin
Number analyzed (Participants) | 47 | 37 | 24 | 20
ng/mL
  Baseline | 5.956 (5.616) | 32.097 (13.624) | 33.917 (15.207) | 32.215 (17.027)
  Tanner 4 | 5.964 (4.582) | 36.867 (20.519) | 44.036 (19.121) | 29.791 (21.892)
  Tanner 5 | 8.338 (7.088) | 38.155 (21.061) | 47.642 (21.269) | 31.182 (20.982)
  Post-Puberty | NA (NA) — Not Measured | NA (NA) — Not Measured | 53.200 (41.323) | 48.445 (31.855)

18. Secondary Outcome: Percent Body Fat
Description: % body fat measured by DXA at time points below
Time Frame: as for outcome 5
Population: 24 participants analyzed in the Obese NT Placebo group are also analyzed in the Obese Placebo group.
Measure: Mean (Standard Deviation); unit: percentage of body fat
Arm/Group | Normal Weight | Obese - NT/Placebo | Obese - Placebo | Obese - Metformin
Number analyzed (Participants) | 47 | 37 | 24 | 20
percentage of body fat
  Baseline | 24.883 (6.452) | 42.126 (5.259) | 44.700 (3.304) | 43.826 (5.412)
  Tanner 4 | 25.054 (6.159) | 43.380 (3.649) | 44.264 (3.489) | 40.610 (7.906)
  Tanner 5 | 25.500 (7.478) | 42.889 (4.688) | 44.555 (3.692) | 39.964 (6.490)
  Post-Puberty | NA (NA) — Not Measured | NA (NA) — Not Measured | 43.962 (5.701) | 41.418 (5.669)

19. Secondary Outcome: Visceral Adipose
Description: Percent Visceral Fat, Measured in a subset (10 per group) by single slice MRI
Time Frame: Baseline, Tanner (puberty) stage 5-average 2.5 yrs from baseline
Population: Data was not collected for some participants at all visits.
Measure: Mean (Standard Deviation); unit: Percent
Groups:
- Obese - NT/Placebo: Obese by BMI. Mix of untreated and Obese-placebo treated.
Arm/Group | Normal Weight | Obese - NT/Placebo | Obese - Metformin | Obese - Placebo
Number analyzed (Participants) | 12 | 6 | 5 | 6
Percent
  Baseline: number analyzed (Participants) | 11 | 6 | 4 | 6
  Baseline | 7.647 (3.702) | 12.007 (2.263) | 12.076 (3.968) | 12.007 (2.263)
  Tanner 5 | 6.322 (2.676) | 12.236 (1.564) | 10.079 (1.886) | 12.236 (1.564)

20. Secondary Outcome: Liver Adipose
Description: Liver fat percent. Measured in a subset (10 per group) by fast MRI technique
Time Frame: Baseline, Tanner (puberty) stage 5-average 2.5 yrs from baseline
Population: Data was not collected for some participants at all visits.
Measure: Mean (Standard Deviation); unit: percentage of liver mass
Groups:
- Obese NT/Placebo: Obese by BMI. Mix of untreated and Obese-placebo treated.
Arm/Group | Normal Weight | Obese NT/Placebo | Obese - Metformin | Obese - Placebo
Number analyzed (Participants) | 12 | 6 | 5 | 6
percentage of liver mass
  Baseline: number analyzed (Participants) | 11 | 6 | 4 | 6
  Baseline | 1.376 (0.594) | 8.290 (7.177) | 13.765 (5.457) | 8.290 (7.177)
  Tanner 5 | 2.208 (0.637) | 8.219 (5.757) | 10.327 (8.023) | 8.291 (5.757)

21. Secondary Outcome: High Density Lipoprotein
Description: Please see primary outcome for more detail about timing of measurement.
Time Frame: as for outcome 1
Population: 24 participants analyzed in the Obese NT Placebo group are also analyzed in the Obese Placebo group.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Normal Weight | Obese - NT/Placebo | Obese - Placebo | Obese - Metformin
Number analyzed (Participants) | 47 | 37 | 24 | 20
mg/dL
  Baseline | 51.442 (8.921) | 39.306 (6.511) | 38.917 (7.003) | 41.368 (7.274)
  Tanner 4 | 51.667 (11.734) | 39.455 (9.533) | 39.455 (9.533) | 42.273 (4.735)
  Tanner 5 | 46.909 (8.498) | 38.944 (8.755) | 39.333 (8.897) | 43.000 (5.916)
  Post-Puberty | NA (NA) — Not Measured | NA (NA) — Not Measured | 40.923 (8.645) | 41.818 (8.171)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at each med visit approximately every 6 months
Groups:
- Obese - Metformin: Dosage form: Metformin 1000 mg tablets Dosage: 1000 mg by mouth twice daily Duration: From early puberty (Tanner 3-4) until puberty completion (Tanner 5), approximately 3 years
  Metformin: After randomization, the study drug (metformin or placebo) is gradually titrated to full dose of 1000 mg BID (or to maximum tolerated, at least 500 mg BID) over a period of 4 weeks to minimize adverse gastrointestinal effects. Participants are seen every three months to measure compliance and dispense new study drug. Every 6 months, they also have a physical examination in order to determine puberty staging. Study measurements (IVGTT, bloodwork, DXA) are performed at Tanner 4 puberty and Tanner 5 (puberty completion), at which time the study drug is stopped. Study measurements will be performed again 6 months after study drug is completed to assess if effects are persistent after study drug is stopped. During the treatment period, all participants receive standard lifestyle counseling.
- Normal Weight (No Treatment): Normal Weight by BMI. No treatment.
- Obese (No Treatment): Obese by BMI. These participants were not prescribed any intervention (Non-treated).
Arm/Group | Obese - Metformin | Obese - Placebo | Normal Weight (No Treatment) | Obese (No Treatment)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/24 | 0/47 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/24 | 0/47 | 0/13
Other Adverse Events (participants affected / at risk) | 11/20 | 14/24 | 0/47 | 0/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Obese - Metformin (N=20) | Obese - Placebo (N=24) | Normal Weight (No Treatment) (N=47) | Obese (No Treatment) (N=13)
Bloating (Gastrointestinal disorders) | 7 | 7 | 0 | 0
Nausea (Gastrointestinal disorders) | 7 | 11 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 6 | 10 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-25): https://cdn.clinicaltrials.gov/large-docs/13/NCT01775813/Prot_SAP_000.pdf